CLINICAL TRIAL: NCT03977675
Title: The Role of HNKs in the Antidepressant Effect of Ketamine
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: PI left the institution
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: NYSPI 7558
Record Dates: First submitted 2019-06-05; First posted 2019-06-06 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Major Depressive Disorder
Keywords: Magnetic Resonance Spectroscopy; Ketamine
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Ketamine 0.3 mg/kg (Experimental): Subjects are assigned to receive a dose of 0.3 mg/kg of Ketamine.
  Interventions: Drug: Ketamine
- Ketamine 0.5 mg/kg (Experimental): Subjects are assigned to receive a dose of 0.5 mg/kg of Ketamine.
  Interventions: Drug: Ketamine
- Ketamine 0.7 mg/kg (Experimental): Subjects are assigned to receive a dose of 0.7 mg/kg of Ketamine.
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — Patients are assigned to one of three ketamine doses (0.3, 0.5, or 0.7 mg/kg) that will be administered intravenously.

SUMMARY:
The objective of the proposed study is to examine the relationship between serum concentrations of HNK and changes in the Hamilton Depression Rating Scale (HDRS), Beck Depression Inventory (BDI), and the Profile of Mood States (POMS), as well as glutamatergic/GABAergic response. To achieve these aims the investigators propose a double-blind, uncontrolled (no placebo, no healthy control subjects) study with several different doses of ketamine. The investigators will conduct MRI scans to measure Glu and GABA before and during the ketamine treatment.

DETAILED DESCRIPTION:
Major depressive disorder (MDD) is a common illness, affecting over 14 million American adults each year. MDD is a leading cause of disability worldwide and is responsible for huge workplace and healthcare costs. The several week delay between onset of treatment and improvement in MDD symptoms with currently available treatments further increases the burden of the disorder. Shortening this delay is a major unmet challenge in the treatment of MDD. Studies report that a single intravenous low dose of a drug called ketamine can bring about substantial improvement in depression in hours, even in patients that have not improved with other antidepressant treatments. Certain aspects of ketamine's drug action are fairly well understood, but the question remains of how these properties relate to antidepressant effect.

Preliminary data support the rapid antidepressant benefit from ketamine but do not show a relationship between clinical improvement and the amount of ketamine, norketamine or dehydronorketamine (DHNK)(two of ketamine's metabolites) in the blood. The investigators hypothesize that a different metabolite of ketamine, hydroxynorketamine (HNK), produces the antidepressant effect of ketamine. The investigators have also used a scanner to measure the effects of ketamine on two major brain chemical transmitters and found that it causes a significant increase (more than 60%) in glutamate (Glu) and gamma aminobutyric acid (GABA) levels in the front of the brain. The investigators hypothesize that this increase in Glu and GABA levels is responsible for the antidepressant action of the drug. Knowing how ketamine works could help to develop better medications that can be used orally and used for maintenance of the improvement seen with ketamine.

ELIGIBILITY:
Inclusion Criteria:

* Current major depressive episode (MDE) as part of major depressive disorder (MDD). May be psychiatric medication-free or, if on psychiatric medications, not responding adequately.
* Off all psychotropic and other types of drugs likely to interact with glutamate for at least 14 days before starting the study OR likely able to tolerate a medication washout.
* Female subjects of child-bearing potential must be using an acceptable method of birth control throughout the study.

Exclusion Criteria:

* Lifetime history of schizophrenia, schizoaffective illness, bipolar disorder, or psychosis.
* First-degree relative with schizophrenia, schizoaffective disorder, or bipolar disorder if the subject is less than 33 years old.
* Significant uncontrolled physical illness.
* Electroconvulsive therapy (ECT) within the last 3 months for current MDE.
* Pregnancy or plans to conceive during the course of study participation.
* Heart pacemaker, body implant or other metal in body.
* Neurological disease or prior head trauma with evidence of cognitive impairment.
* Claustrophobia sufficient to preclude MRI.
* Prior ineffective trial of, or adverse effect to, ketamine.
* IV drug use or history of ketamine use as a recreational drug ≥ 2 times or an adverse reaction to ketamine; any other drug or alcohol dependence within past 6 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2020-07-02 (Actual); Study Completion 2020-07-02 (Actual)

PRIMARY OUTCOMES:
Change in HNK Plasma Concentration | Baseline and 80 minutes post-infusion
  HNK levels will be measured after ketamine administration.
Change in DHNK Plasma Concentration | Baseline and 80 minutes post-infusion
  DHNK levels will be measured after ketamine administration.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Grunebaum, MD, Principal Investigator — New York Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No